CLINICAL TRIAL: NCT02087774
Title: The Effects of a Brief Physical Activity Program on Elementary School Students' Physical Fitness
Brief Title: Brief Physical Activity Program to Increase Physical Fitness in Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Rebecca Hayes, Resident Physician, Marshall University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 498505-2
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control School (No Intervention): Control School received no intervention.
- 6 minutes activity (Experimental): Implementation of 6 minutes of physical activity daily into the school day routine. Children can jog in place, do jumping jacks or dance.
  Interventions: Behavioral: 6 minutes activity

INTERVENTIONS:
Behavioral: 6 minutes activity — Group added 6 minutes of physical activity daily during school day.
  Arms: 6 minutes activity

SUMMARY:
The investigators hypothesized that the addition of 6 minutes of exercise during the school day would increase physical fitness in elementary school students as demonstrated by longer distances run in 2 minutes and a decrease in heart rate at the end of the exercise.

DETAILED DESCRIPTION:
Intervention group played music for 6 minutes each morning in addition to recess and physical activity classes. Baseline fitness data and after-intervention data were compared.

ELIGIBILITY:
Inclusion Criteria:

* All students were invited to participate.

Exclusion Criteria:

* Lack of parental consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca H Hayes, M.D., Principal Investigator — Marshall University
Locations (1):
- Marshall University, Huntington, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Two schools participated in the intervention which consisted on 6 minutes of exercise a day and incentives like pedometers and physical fitness prizes.
  One intervention school implemented the program with responsibility given to the principal (school-wide group) and the other school asked the individual teachers to implement the program daily (classroom based group).
  Physical Activity and Incentives
Period: Overall Study
Arm/Group | Control School | Intervention Group
Started | 150 | 150
Completed | 142 | 130
Not Completed | 8 | 20
Not completed — Were absent day of data collection | 8 | 20

BASELINE CHARACTERISTICS:
Population: Both groups were located in a rural, eastern state within 75 miles from one another
Groups:
- Intervention Group: Oneparticipated in the intervention which consisted on 6 minutes of exercise a day and incentives like pedometers and physical fitness prizes.
  The responsibility was given to the principal to implement the program.
  Physical Activity and Incentives
- Total: Total of all reporting groups
Arm/Group | Control School | Intervention Group | Total
Number analyzed (Participants) | 142 | 130 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 142 | 130 | 272
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 71 | 125
  Male | 88 | 59 | 147
Region of Enrollment [Number; unit: participants]
  United States | 142 | 130 | 272
Grade level [Mean (Standard Deviation); unit: grade] | 3.1 (1.4) | 2.9 (1.4) | 3.0 (1.4)
75 foot laps completed [Mean (Standard Deviation); unit: laps completed] | 13.5 (1.9) | 13 (2) | 13.3 (2)
After exercise- heart rate [Mean (Standard Deviation); unit: beats per minute] | 163 (27.9) | 164.8 (23.8) | 163.9 (25.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to After Intervention in 75 Foot Laps Completed in 2 Minutes
Description: Subjects run for 2 minutes around cone separated by 75ft. One lap was one 75 foot length completed.
  Difference in laps completed from baseline was taken.
Time Frame: Baseline to 12 weeks later
Measure: Mean (95% Confidence Interval); unit: Difference in Laps Completed
Arm/Group | Control School | Intervention Group
Number analyzed (Participants) | 142 | 130
Difference in Laps Completed | -0.08 (Referent) [-0.10 to -0.04] | 0.53 [0.17 to 1.1]

2. Primary Outcome: Change From Baseline to After Intervention for After-Exercise Heart Rate
Description: Immediate cool-down, after-exercise heart rate was taken.
  Difference in heart rate from baseline measurements is reported
Time Frame: Baseline to 12 weeks later
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Control School | Intervention Group
Number analyzed (Participants) | 142 | 130
beats per minute | 16.0 [10.5 to 20.3] | -21.4 [-29.1 to -14.5]

ADVERSE EVENTS:
Time Frame: Immediately and for 3 months after
Arm/Group | Control School | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/130
Other Adverse Events (participants affected / at risk) | 0/142 | 0/130

LIMITATIONS AND CAVEATS:
Non-randomized, controlled design. Majority of subject were caucasian, from Appalachian region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes